CLINICAL TRIAL: NCT00899483
Title: Can Enhanced Glycaemic Control in Type II Diabetics Improve Myocardial Protection During Coronary Artery Bypass Grafting?
Brief Title: Can Enhanced Glycemic Control in Type II Diabetics Improve Myocardial Protection During Coronary Artery Bypass Grafting?
Acronym: GUIDE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital Birmingham (Other)
Collaborators: British Heart Foundation (Other)
Responsible Party: Professor Robert S Bonser, University Hospital Birmingham
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RRK3545
Record Dates: First submitted 2009-05-11; First posted 2009-05-12 (Estimated); Last update posted 2009-05-12 (Estimated); Status verified 2009-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — glucose-insulin-potassium cardioplegic solution

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Administered with glucose potassium insulin solution to achieve euglycaemia 4.0-6.0 mmol/L
  Interventions: Drug: Glucose potassium insulin solution
- 2 (No Intervention): Normal departmental practice using dextrose insulin infusion

INTERVENTIONS:
Drug: Glucose potassium insulin solution — Enhanced glycaemic control in diabetics with glucose-potassium-insulin solution
  Arms: 1

SUMMARY:
The investigators have previously demonstrated that the administration of insulin in the form of an infusion with additional sugar and potassium may improve cardiovascular performance and reduce biochemical evidence of heart muscle injury in non-diabetic patients undergoing coronary artery surgery. The investigators now seek to demonstrate that similar benefits can be achieved in diabetic patients by administering insulin to maintain as near absolutely normal sugar levels as possible.

ELIGIBILITY:
Inclusion Criteria:

* Type II diabetes mellitus patients (as defined by WHO)
* Diet, oral hypoglycaemic or insulin therapy
* Undergoing elective and urgent coronary artery bypass surgery

Exclusion Criteria:

* Non-diabetics
* Emergency and redo CABG
* < 18 years
* Pregnancy
* Dialysis-dependence
* History of CVA/TIA < 6 months
* Heart valve disease requiring surgery
* STEMI < 3 months

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-07; Primary Completion 2012-07 (Estimated)

PRIMARY OUTCOMES:
The difference in the mean left ventricular end-systolic volume index (LVESVI) after CABG and the amount of new permanent injury detected in the late CMRI study | 3 months post CABG

SECONDARY OUTCOMES:
Glycaemic control will be assessed 2 hours pre-operatively and 72 hours post-operatively. Measurement timings will be standardized allowing comparison of glycaemic control during different time-periods. | 72 hours post CABG

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Birmingham, Birmingham, West Midlands, United Kingdom

REFERENCES:
- [Derived] Bellon F, Sola I, Gimenez-Perez G, Hernandez M, Metzendorf MI, Rubinat E, Mauricio D. Perioperative glycaemic control for people with diabetes undergoing surgery. Cochrane Database Syst Rev. 2023 Aug 1;8(8):CD007315. doi: 10.1002/14651858.CD007315.pub3. PMID 37526194